CLINICAL TRIAL: NCT05929547
Title: An In Depth Study Examining Patterns in the Clinical Trial Experiences of Squamous Cell Carcinoma Patients
Brief Title: Patient Perspectives in Squamous Cell Carcinoma Clinical Trials
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 80490767
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Squamous Cell Carcinoma
Keywords: squamous cell carcinoma
MeSH Terms: conditions — Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical research participation has historically been heavily biased toward specific demographics.

This study will invite several participants to gather a wide range of information on clinical trial experiences for squamous cell carcinoma patients. The aim of the study is to identify the factors that limit the ability of a person to enroll in, as well as complete a clinical trial for treatment of squamous cell carcinoma.

People with squamous cell carcinoma who are invited to take part in clinical research will benefit from the analysis of the data.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old
* Confirmed diagnosis of squamous cell carcinoma
* Subjects willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examination.

Exclusion Criteria:

* Inability to provide written informed consent
* Is pregnant, breastfeeding or expecting to conceive within the projected duration of the study
* Enrolled in another research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with squamous cell carcinoma who are actively considering enrolling in a clinical trial for said condition, but have not yet completed enrollment and randomization phases.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to enroll in a squamous cell carcinoma clinical trial | 3 months
Rate of patients who remain in squamous cell carcinoma clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Leis M, Singh A, Li C, Ahluwalia R, Fleming P, Lynde CW. Risk of Vulvar Squamous Cell Carcinoma in Lichen Sclerosus and Lichen Planus: A Systematic Review. J Obstet Gynaecol Can. 2022 Feb;44(2):182-192. doi: 10.1016/j.jogc.2021.09.023. Epub 2021 Oct 19. PMID 34678521
- [Background] Gupta S, Kamboj M, Narwal A. Knowing the unknown in oral squamous cell carcinoma: An observational study. J Cancer Res Ther. 2020 Apr-Jun;16(3):494-499. doi: 10.4103/jcrt.JCRT_898_18. PMID 32719256
- [Background] Schlessinger DI, Iyengar S, Yanes AF, Chiren SG, Godinez-Puig V, Chen BR, Kurta AO, Schmitt J, Deckert S, Furlan KC, Poon E, Cartee TV, Maher IA, Alam M, Sobanko JF. Development of a core outcome set for clinical trials in squamous cell carcinoma: study protocol for a systematic review of the literature and identification of a core outcome set using a Delphi survey. Trials. 2017 Jul 12;18(1):321. doi: 10.1186/s13063-017-2069-2. PMID 28701207

DOCUMENTS (1):
  • Informed Consent Form (2023-06-23): https://cdn.clinicaltrials.gov/large-docs/47/NCT05929547/ICF_000.pdf